CLINICAL TRIAL: NCT00928148
Title: A Phase 2, Randomized, Double-Blind, Multi-Center, Placebo- and Active-Controlled, Crossover Study of SPD465 in Adults With Attention-Deficit Hyperactivity Disorder
Brief Title: The Safety and Efficacy of SPD465 in Adults With Attention Deficit Hyperactivity Disorder (ADHD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: SPD465-201
Record Dates: First submitted 2009-06-23; First posted 2009-06-25 (Estimated); Last update posted 2021-06-03 (Actual); Status verified 2021-05

CONDITIONS: Attention-Deficit/Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- SPD465 (50 or 75 mg) (Experimental)
  Interventions: Drug: SPD465
- Immediate Release Amphetamine salt (25 mg) (Active Comparator)
  Interventions: Drug: Immediate Release Amphetamine Salt
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SPD465 — 50 or 75 mg once daily for 7 days
  Arms: SPD465 (50 or 75 mg)
Drug: Immediate Release Amphetamine Salt — 25 mg once daily for 7 days
  Arms: Immediate Release Amphetamine salt (25 mg)
Drug: Placebo — Once daily for 7 days
  Arms: Placebo

SUMMARY:
This is a phase 2, randomized, multi-center, double-blind, 3-period and 3-treatment crossover study designed to evaluate the safety and duration of efficacy of SPD465 (50 or 75 mg) compared with placebo and an immediate release amphetamine salt formulation (25 mg) in adults with ADHD. The controlled environment used in this study is an analog classroom setting adapted for a 16-hour adult day.

ELIGIBILITY:
Inclusion Criteria:

* Adult men and non-pregnant women between the ages of 18 and 55
* Confirmed diagnosis of ADHD as defined by the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, Text Revision (DSM-IV-TR)
* Baseline ADHD score of at least 24

Exclusion Criteria:

* Weight less than 100 pounds or greater than 250 pounds
* Psychiatric diagnosis such as a severe comorbid Axis II or Axis I disorder
* Pregnancy or breastfeeding
* History of seizures
* Positive urine drug screen

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 86 (Actual)
Dates: Start 2004-06-14 (Actual); Primary Completion 2004-11-20 (Actual); Study Completion 2004-11-20 (Actual)

PRIMARY OUTCOMES:
To assess the duration of efficacy of SPD465 compared to placebo and immediate release amphetamine formulation in adults with ADHD using the Permanent Product Measure of Performance (PERMP) math test | -0.5, 2, 4, 8, 12, 14 and 18 hours post-dose

SECONDARY OUTCOMES:
To assess the duration of efficacy of SPD465 compared with placebo and immediate release amphetamine on ADHD symptoms as determined by the ADHD-rating scale (ADHD-RS) | 5, 10 and 15 hours post-dose
To assess the duration of efficacy of SPD465 compared with placebo and immediate release amphetamine on ADHD symptoms as determined by the Swanson, Kotkin, Agler, M. Flynn, and Pelham (SKAMP) scale | 5, 10, and 15 hours post-dose
To assess the impact of SPD465 compared with placebo and immediate release amphetamine on sleep as measured by the modified Pittsburgh Sleep Quality Index (PSQI) | 21 days
To evaluate the safety of SPD465 based on occurrence of treatment-emergent adverse events (TEAEs), blood pressure (BP), heart rate, electrocardiogram (ECG), and clinical laboratory findings | 21 days

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda

REFERENCES:
- [Derived] Wigal T, Brams M, Frick G, Yan B, Madhoo M. A randomized, double-blind study of SHP465 mixed amphetamine salts extended-release in adults with ADHD using a simulated adult workplace design. Postgrad Med. 2018 Jun;130(5):481-493. doi: 10.1080/00325481.2018.1481712. Epub 2018 Jun 18. PMID 29809075